CLINICAL TRIAL: NCT00719459
Title: A Randomized, Open-Label, Single-Dose, Parallel-Design, Bioequivalence Study of Hospira Iron Sucrose Injection Compared to Venofer® Injection USP in Healthy Subjects.
Brief Title: Bioequivalency Study Comparing Hospira's Generic Iron Sucrose Injection to Venofer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRON-07-04
Record Dates: First submitted 2008-07-15; First posted 2008-07-21 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2015-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Hospira Iron Sucrose
  Interventions: Drug: Iron Sucrose
- 2 (Active Comparator): Venofer
  Interventions: Drug: Iron Sucrose

INTERVENTIONS:
Drug: Iron Sucrose — Venofer 20 mg/mL
  Arms: 2
Drug: Iron Sucrose — Iron sucrose 20 mg/mL
  Arms: 1

SUMMARY:
The primary objective of this study is to assess the bioequivalence of the test product Hospira Iron Sucrose 20 mg/mL (Hospira, Inc.) to the reference product Venofer® 20 mg/mL following intravenous administration to healthy subjects.

DETAILED DESCRIPTION:
Iron is essential to the synthesis of hemoglobin (Hb) to maintain oxygen transport and to the function and formation of other physiologically important heme and nonheme compounds. Iron deficiency may be caused by blood loss during dialysis, increased erythropoiesis following administration of epoetin, and insufficient absorption of iron from the gastro-intestinal tract. Most dialysis patients require intravenous iron supplementation to replenish iron stores.

Iron sucrose is used to replenish body iron stores in patients with iron deficiency on chronic hemodialysis and receiving erythropoietin. In these patients iron deficiency is caused by blood loss during dialysis procedure, increased erythropoiesis, and insufficient absorption of iron from the gastrointestinal tract. Most hemodialysis patients require intravenous iron to maintain sufficient iron stores to achieve and maintain a hemoglobin level of 11-12 g/dL.

Subjects who fulfill the inclusion/exclusion criteria after screening will be randomized to receive 100 mg of iron sucrose as either Hospira Iron Sucrose or Venofer®.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers between 18 and 55 years of age (both inclusive).
2. Having a Body Mass Index (BMI) between 18.5 and 32.0 kg/m2 (both inclusive).
3. If female, subject must be either postmenopausal for at least 1 year, surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or practicing birth control:

   * hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration
   * intrauterine device (IUD)
   * double-barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream).

   If hormonal contraceptives are used, the specific contraceptive must have been used for at least 3 months prior to study drug administration. If the subject is currently using a hormonal contraceptive, she should also use a barrier method during this study and for 1 month after study completion.
4. Must have, in the investigator's opinion, no abnormal laboratory evaluations taken at Screening visit or admission to the Phase 1 unit on Day -1.
5. Must be a non-smoker (defined as a subject who has not smoked for 3 months) and agree to abstain from alcohol for 24 hours prior to each dosing treatment and while a resident in the treatment unit.
6. Able to provide written informed consent after risks and benefits of the study have been explained.
7. Able to communicate effectively with study personnel.

Exclusion Criteria:

1. Documented bleeding disorders, acute bleeding or recently documented hemorrhage.
2. Any disease or condition that might interfere with the absorption, distribution, metabolism, or excretion of the study drug or would place the subject at increased risk.
3. History of drug abuse or alcohol abuse within 2 years of study enrollment as determined by the investigator or a positive urine drug test prior to Day -1.
4. Use of any prescription medicine within 14 days prior to start of the study, or over the counter medications or herbal remedies within 3 days prior to study entry (vitamins or calcium supplements allowed, except iron supplements).
5. Use of iron supplements within 3 months of the start of the study.
6. A subject with anemia (hemoglobin < 8 mg/dL).
7. Relative or absolute iron deficiency or iron overload.
8. Clinically significant medical or psychiatric illness currently or within 30 days of study entry as determined by investigator.
9. Significant drug sensitivity or a significant allergic reaction to any drug.
10. Known hypersensitivity or idiosyncratic reaction to iron sucrose injection or any other related drugs.
11. A positive result at screening for HIV, Hepatitis B or C.
12. A subject who has been administered an injectable drug within 14 days prior to the start of the study.
13. A subject who has donated or lost 475 mL (i.e., 1 pint) or more blood volume (including plasmaphoresis) or had a transfusion of any blood product within 3 months prior to the initial study drug administration.
14. Current participation or participation within 30 days prior to the initial study drug administration in a drug or other investigational research study.
15. A subject who may not be able to comply with the safety monitoring requirements of this clinical trial or is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07-13 (Actual)

PRIMARY OUTCOMES:
Bioequivalence - Assessed by constructing the 90% confidence interval (CI) for the geometric mean test/reference ratios of Cmax for both baseline-adjusted total iron and baseline-adjusted transferrin-bound iron | Pharmacokinetic sampling at pre-dose (15, 10 and 5 minutes) and Post-dose 5, 10, 20, 30, 45 minutes, and 1.0,2.0,3.0,4.0,6.0,8.0, 12.0, 14.0, and 24.0 hours.
  Test: Hospira Iron Sucrose Injection; Reference: Venofer Injection
Bioequivalence - Assessed by constructing the 90% CI for the geometric mean test/reference ratios of AUC0-t for both baseline-adjusted total iron and baseline-adjusted transferrin-bound iron | Pharmacokinetic sampling at pre-dose (15, 10 and 5 minutes) and Post-dose 5, 10, 20, 30, 45 minutes, and 1.0,2.0,3.0,4.0,6.0,8.0, 12.0, 14.0, and 24.0 hours.
  Test: Hospira Iron Sucrose Injection; Reference: Venofer Injection

SECONDARY OUTCOMES:
Time of maximum concentration (Tmax) for baseline-adjusted total iron and baseline-adjusted transferrin-bound iron | Pharmacokinetic sampling at pre-dose (15, 10 and 5 minutes) and Post-dose 5, 10, 20, 30, 45 minutes, and 1.0,2.0,3.0,4.0,6.0,8.0, 12.0, 14.0, and 24.0 hours.
Half life (t1/2) for baseline-adjusted total iron and baseline-adjusted transferrin-bound iron | Pharmacokinetic sampling at pre-dose (15, 10 and 5 minutes) and Post-dose 5, 10, 20, 30, 45 minutes, and 1.0,2.0,3.0,4.0,6.0,8.0, 12.0, 14.0, and 24.0 hours.
Elimination rate constant (λz) for baseline-adjusted total iron and baseline-adjusted transferrin-bound iron | Pharmacokinetic sampling at pre-dose (15, 10 and 5 minutes) and Post-dose 5, 10, 20, 30, 45 minutes, and 1.0,2.0,3.0,4.0,6.0,8.0, 12.0, 14.0, and 24.0 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Bio-Kinetic Clinical Applications, Springfield, Missouri, United States